CLINICAL TRIAL: NCT01981382
Title: Characterizing Pain Sensitivity in Persistent Nonspecific Low Back Pain
Brief Title: Characterizing the Role of Pain Sensitivity in Acute to Persistent Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01NR013932-01 (NIH); R01NR013932-01 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
Keywords: low back pain; pain sensitivity; genes; gene expression,; quantitative sensory testing
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Incident cases: Persistent nonspecific low back pain
- Controls: Acute low back pain that resolves in <6 months

SUMMARY:
This research study will examine whether enhanced pain sensitivity increases the risk of persistent low back pain. The study will address the highly prevalent and costly condition of persistent low back pain and a major obstacle for the implementation of clinical strategies to improve patient outcomes. The knowledge gained from this study may lead to a better understanding of the biological mechanisms that contribute to persistent low back pain and will inform future work to develop predictive measures of persistent low back pain risk, evaluative measures to examine treatment efficacy, and possibly biomarker assay(s) to identify patients who are at increased risk of persistent low back pain.

DETAILED DESCRIPTION:
The specific aims (SA) of the proposed study are to:

Specific Aim 1. Characterize (A) the differences in pain sensitivity between incident cases and controls at low back pain onset and (B) changes in pain sensitivity over time in incident cases.

H1.A Incident cases will have increased pain sensitivity compared with controls at low back pain onset.

H1.B Incident cases will have increased pain sensitivity over time.

Specific Aim 2. Compare (A) genetic polymorphisms at low back pain onset between incident cases and controls and mRNA expression of candidate genes at LBP onset and at 6 weeks between incident cases and controls; and (B) differential expression levels of candidate genes over time in incident cases.

H2.A Incident cases will have a higher frequency of polymorphisms and differential expression levels of candidate genes at low back pain onset compared with controls.

H2.B Examine expression levels of candidate genes over time in incident cases.

Specific Aim 3. Determine the contribution of enhanced pain sensitivity, cofactors (clinical/psychosocial/environmental), genetic polymorphisms, and mRNA expression of candidate genes on the risk of persistent low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years of age;
2. diagnosed with an acute episode of nonspecific LBP present for >24 hours but <4 weeks duration and preceded by at least 1 pain-free month; and
3. comprehend English

Exclusion Criteria:

1. <18 or >50 years of age;
2. chronic pain at another site or associated with a painful condition (eg., fibromyalgia, neuropathy, rheumatoid arthritis);
3. previous spinal surgery;
4. presence of neurological deficits;
5. history of comorbidities that affect sensorimotor function (eg., multiple sclerosis, spinal cord injury, diabetes); and
6. untreated psychological disorders (major depression, bipolar disorder, schizophrenia)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women between the ages of 18-50 years of age who are diagnosed with an acute nonspecific LBP episode defined as pain anywhere in the region of the low back bound superiorly by T12 and inferiorly by the buttock crease, which has been present for >24 hours but <4 weeks duration and was preceded by at least 1 pain-free month.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Experimental Pain Threshold | 6 months
  Quantitative sensory testing will be used to evaluate pain sensitivity over time

SECONDARY OUTCOMES:
mRNA expression of pain sensitivity genes | 6 months
  Expression of pain sensitivity genes will be measured over time

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Starkweather, PhD, RN, Principal Investigator — University of Connecticut School of Nursing

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon completion of study and final acceptance of publications

REFERENCES:
- [Result] Starkweather AR, Lyon DE, Kinser P, Heineman A, Sturgill JL, Deng X, Siangphoe U, Elswick RK, Greenspan J, Dorsey SG. Comparison of Low Back Pain Recovery and Persistence: A Descriptive Study of Characteristics at Pain Onset. Biol Res Nurs. 2016 Jul;18(4):401-10. doi: 10.1177/1099800416631819. Epub 2016 Feb 16. PMID 26883808
- [Result] Starkweather AR, Ramesh D, Lyon DE, Siangphoe U, Deng X, Sturgill J, Heineman A, Elswick RK Jr, Dorsey SG, Greenspan J. Acute Low Back Pain: Differential Somatosensory Function and Gene Expression Compared With Healthy No-Pain Controls. Clin J Pain. 2016 Nov;32(11):933-939. doi: 10.1097/AJP.0000000000000347. PMID 26736025